CLINICAL TRIAL: NCT02759276
Title: Inflammatory Biomarkers and Endothelial Function Assessed by Venous Occlusion Plethysmography and Nailfold Videocapillaroscopy in Patients With Resistant Hypertension, Stages 1 and 2 and Normotensive
Brief Title: Microcirculation and Inflammatory Markers in Patients With Resistant, Stages 1/2 Hypertension and Normal Blood Pressure
Acronym: MICRORAH
Status: Completed | Type: Observational
Sponsor: Daniel Alexandre Bottino (Other)
Collaborators: Rio de Janeiro State University (Other)
Responsible Party: Sponsor-Investigator, Daniel Alexandre Bottino, M.D., PhD, Rio de Janeiro State University
Organization: Rio de Janeiro State University (Other)
Other Study IDs: RiodeJaneiro_StateUniversity; BIOVASC-UERJ (Other: Clinical and Experimental Research Lab on Vascular Biology)
Record Dates: First submitted 2016-04-20; First posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: High Blood Pressure
Keywords: Nailfold Videocapillaroscopy; Venous Occlusion Plethysmography; Endothelial Function; Microcirculation; Inflammatory Biomarkers
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Resistant Hypertension (RH): uncontrolled hypertension, with values ≥140/90 mmHg, using three or more antihypertensive drugs of different classes, including a diuretic, or controlled hypertension with four or more drugs.
- Stages 1 and 2 Hypertension (MMH): According to the VI Brazilian Guidelines of hypertension, with blood pressure levels ranging from 140/90 mmHg to 179/109 mmHg, with up to two antihypertensive drugs of different classes and blood pressure levels controlled in the last two months.
- Normotensive (CG): Blood Pressure <140/90 mmHg and without comorbidities.

SUMMARY:
Nailfold videocapillaroscopy (NVC), Venous occlusion Plethysmography (VOP) and inflammatory biomarkers have been used to study endothelial function in patients with resistant hypertension, stages 1 and 2 hypertension and normotensive. This was a cross-sectional study.

DETAILED DESCRIPTION:
Microcirculation determines peripheral resistance contributing to increased blood pressure. The nailfold videocapillaroscopy (NVC), Venous occlusion Plethysmography (VOP) and biomarkers can be used to evaluate the microcirculation in arterial hypertension (AH). The objective of this study is to analyze the behavior of serum inflammatory markers and study the microcirculation by nailfold videocapillaroscopy (NVC) and Venous Occlusion Plethysmography in patients with resistant hypertension (RH), with stages 1 and 2 hypertension (MMH ) and normotensive (CG). A cross-sectional study with 75 patients has been performed: 25 with resistant hypertension (RH), 25 with stages 1 and 2 hypertension (MMH) and 25 normotensive (CG). All underwent anamnesis, dosage serum markers and conducting NVC, VOP. Hypertensive patients without statin use and with controlled or uncontrolled blood pressure were also analyzed. For the statistical analysis were used: Kruskal -Wallis ANOVA, Dunn test and ANCOVA for correction of confusion factors such as age and BMI.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of controlled High Blood Pressure stages 1 and 2 (blood pressure levels from 140/90 mmHg to 179/109 mmHg) .
* Resistant Hypertension (uncontrolled hypertension, with values ≥140/90 mmHg, using three or more antihypertensive drugs of different classes, including a diuretic, or controlled hypertension with four or more drugs).
* Normal Blood Pressure.

Exclusion Criteria:

* Diabetes Mellitus, Types 1 or 2.
* Heart Failure.
* Myocardial infarction or stroke with less than three months of the event.
* Chronic kidney disease.
* Use of hormonal or non-hormonal anti-inflammatory drugs.
* Recent trauma (less than three months).
* Autoimmune diseases.
* Infectious processes in activity.
* Neoplasia.
* Aspirin use (anti-inflammatory dose).
* Obesity grade III (Body Mass Index>40 kg/m2).

Ages: 27 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First Day: Full clinical examination was performed, including measurements of at-rest blood pressure, weight and height in order to calculate Body Mass Index (BMI), waist and hip measurements.
  Second Day: drawing blood for laboratory analyses, Nailfold Videocapillaroscopy and Venous Occlusion Plethysmography.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Blood Pressure (mmHg) | 1 day
  Hemodynamic Variable

SECONDARY OUTCOMES:
Functional Capillary Density (FCD, number capillaries/mm2 ) | 1 day
  Microcirculatory variable from Nailfold Videocapillaroscopy
Afferent Capillary Diameter (micrometer) | 1 day
  Microcirculatory variable from Nailfold Videocapillaroscopy
Apical Capillary Diameter (micrometer) | 1 day
  Microcirculatory variable from Nailfold Videocapillaroscopy
Efferent Capillary Diameter (micrometer) | 1 day
  Microcirculatory variable from Nailfold Videocapillaroscopy
Red Blood Cell Velocity (mm/s) | 1 day
  Microcirculatory variable from Nailfold Videocapillaroscopy
Maximum Red Blood Cell Velocity (mm/s) | 1 day
  Microcirculatory variable from Nailfold Videocapillaroscopy
Time to reach Maximum Red Blood Cell Velocity (s) | 1 day
  Microcirculatory variable from Nailfold Videocapillaroscopy
Waist circumference (cm) | 1 day
  Anthropometrical Variable
Hip circumference (cm) | 1 day
  Anthropometrical Variable
Waist to Hip Ratio | 1 day
  Anthropometrical Variable
Body Mass Index (Kg/m2) | 1 day
  Anthropometrical Variable
Maximal Forearm Blood Flow during reactive Hyperemia | 1 day
  Vascular Reactivity Variables from Venous Occlusion Plethysmography
Maximal Forearm Blood Flow after sublingual nitroglycerine | 1 day
  Vascular Reactivity Variables from Venous Occlusion Plethysmography
Vascular Cell Adhesion Molecule (VCAM, ng/dl) | up to 2 weeks
  Inflammatory Biomarker
Intercellular Adhesion Molecule (ICAM, ng/dl) | up to 2 weeks
  Inflammatory Biomarker
Adiponectin (ng/dl) | up to 2 weeks
  Inflammatory Biomarker
Endothelin (pg/dl) | up to 2 weeks
  Inflammatory Biomarker
C Reactive Protein (CRP, mg/dl) | up to 2 weeks
  Inflammatory Biomarker

IPD SHARING:
Plan to Share IPD: No